CLINICAL TRIAL: NCT03279952
Title: Neurophysiological Markers of Pediatric Irritability and Its Response to Intervention
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: challenge in recruitment]
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Raman Baweja, Associate Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB: 00008087
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Central Nervous System Stimulants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- medication arm (Other): CNS Stimulant
  Interventions: Drug: CNS Stimulant

INTERVENTIONS:
Drug: CNS Stimulant — Participants will be stabilized by any FDA approved CNS stimulant medication during open label trial.

SUMMARY:
There has been an increasing focus on the adverse impacts of irritability, defined as increased tendency towards anger. Irritability worsens peer relationships, family functioning, academic performance and is a risk factor for depression, suicide and substance use and is one of the main reasons why children get referred for treatment. It has been identified as transdiagnostic entity meriting investigation as a treatment target for personalized intervention given its prevalence and morbidity. Most children with prominent irritability also meet criteria for Attention Deficit Hyperactivity Disorder (ADHD) but only a subset of children with ADHD manifest impairing levels of irritability. Irritability levels are only minimally correlated with severity of ADHD symptoms suggesting that irritability is not simply a manifestation of severe ADHD. The first line treatment for irritability in children with ADHD is to optimize the dose of the CNS stimulant. However, there is great heterogeneity in response, with baseline mood lability being the best marker for both improving and worsening irritability. In addition, increased irritability is one of the most common reasons why parents stop these medications. The unpredictability in response to CNS stimulants has led to the increasing use of antipsychotics and other non-evidence based treatments for ADHD. It is unknown what drives this heterogeneity in response in part because little is known about the underlying causal mechanisms for irritability in youth with ADHD. Two areas theorized to contribute to irritability include impairments in learning from experience (instrumental learning) and sensitivity to reward and loss.1 There are objective methods for measuring these domains in children through the use of even-related potentials (ERPs)- synchronous neural activity in response to a stimulus. Reward positivity (RewP) is an ERP component occurring in response to feedback on task performance that can be broken down to separate reward and loss components. Irritability is thought to arise due to the combination of an enhanced drive for reward coupled with an excessive response to loss. No prior work has examined associations of RewP with irritability in ADHD. However, abnormalities in RewP and elevated irritability have both been established as risk factors for depression, suggesting that RewP may also predict irritability. Error related negativity (ERN) reflects the preconscious detection of potential conflict serving as an early warning signal for errors. Error detection is one of the first steps for instrumental learning. It is impaired in some youth with ADHD, with a suppressed ERN correlated with reduced error processing. CNS stimulants improve ERN amplitude and impaired error processing. We theorize that abnormalities in RewP and ERN in children with ADHD will serve as respective markers for severity of irritability and subsequent treatment response to CNS stimulants. If successful, we will have identified a causal pathway for irritability that will aide treatment development and identified a reliable biomarker for the current first line treatment for irritability in ADHD (CNS Stimulants), while providing care to a significantly impaired group of local children for whom few evidence-based treatments exist.

DETAILED DESCRIPTION:
There has been an increasing focus on the adverse impacts of irritability, defined as increased tendency towards anger.In children, irritability manifests as a persistently negative mood and frequent temper outbursts. Severe, persistent irritability has been conceptualized as Disruptive Mood Dysregulation Disorder (DMDD) with 3% of children meeting criteria for it. Most youth with DMDD have Attention Deficit Hyperactivity Disorder (ADHD) but only a subset of patients with ADHD exhibit impairing irritability. Even in children not meeting full DMDD criteria, irritability causes a range of impairments and is a risk factor for depression, suicide and substance use. Irritability has been identified as transdiagnostic entity meriting investigation as a target for personalized intervention. Irritability levels are only minimally correlated with severity of ADHD symptoms or impairments in executive functioning, suggesting that irritability is distinct and not simply a manifestation of severe ADHD. Presently, the first line treatment for irritability in children with ADHD is to optimize the dose of the CNS stimulant. However, there is great heterogeneity in response, with some children experiencing complete remission of their irritability and others experience worsening irritability. Increased irritability is one of the most common reasons why parents stop these medications. It is unknown what drives this heterogeneity in response as no reliable treatment markers have been identified. The unpredictability of CNS stimulants has led to the increasing use of atypical antipsychotics for the off label treatment of ADHD. While effective, these medications are associated with concerning side effects.

In order to identify markers of treatment response, it is necessary to delineate the causal pathways underlying irritability. However, the mechanisms driving irritability are largely unknown. Two areas theorized to contribute to irritability are impairments in learning from experience (instrumental learning) and sensitivity to reward and loss. There are objective, reliable methods for measuring these domains in children through the use of event related potentials (ERPs), synchronous neural activity derived from the electroencephalogram (EEG) in response to a stimulus. Reward positivity (RewP) is an ERP occurring in response to feedback on task performance that can be broken down to separately analyze response to gain (delta frequency) and loss (theta frequency). No prior work has examined these components of RewP with irritability but others have found unique associations of each with depression. As irritability is an established risk factor for depression, it is reasonable to surmise that RewP may predict irritability as well. Error related negativity (ERN) reflects the preconscious detection of potential conflict, serving as an early warning signal for errors and a first step to adapting behavior in response to achieve a desired goal (e.g., instrumental learning.) A subset of children with ADHD exhibit a suppressed ERN on cognitive tasks, and ERN amplitude is associated with task performance. When suppressed, CNS stimulants normalize ERN, which is correlated with improved task performance. We theorize that abnormalities in RewP to reward and loss on a monetary guessing task will predict the severity of irritability, while ERN amplitude on a response inhibition task will predict the degree of improvement in irritability after dose optimization of CNS stimulants. These associations will be assessed in 47 children with ADHD and elevated levels of irritability using daily parent ratings gathered before and after optimization of CNS stimulant. To address the great variability in a child's daily behavior, we will use the recommended collection format of ecological momentary assessment (EMA) to gather multiple daily ratings of irritability. Lastly, there is a longstanding concern that CNS stimulants may lead to rebound irritability late in the day as their effects fade. It is unclear if this simply represents a return to the premedication baseline that parents perceive as more severe after observing improved behavior earlier in the day or a true worsening in irritability. Therefore, we will use EMA to compare changes in irritability during medicated times of day versus unmedicated times, theorizing that greater daytime improvement will be associated with parents rating worse evening behavior.

Aim1: Examine the capacity of lab measurements of reward sensitivity to predict irritability in ADHD children H1: After controlling for relevant covariates, gain-related delta and loss-related theta activity in the EEG during a reward-guessing task will each correlate with levels of the child's irritability.

H2:Children with elevated levels of both loss related theta &gain-related delta will exhibit the greatest irritability.

Aim2: Examine the capacity of ERN amplitude during a response inhibition task done in the unmedicated state to predict the capacity of CNS stimulants to reduce irritability in children with ADHD.

H1: Smaller baseline ERN will predict greater improvement in irritability with optimization of stimulant dose.

Aim3: Examine the phenomena of rebound irritability with wear-off of the therapeutic effect of CNS stimulants.

H1: Greater reductions in irritability when the CNS stimulant is active will be associated with parents reporting increasing irritability after the stimulant has worn off.

ELIGIBILITY:
Inclusion Criteria: 1. Ages 5-12: CNS stimulant medications are commonly used and well studies in this age range (Mixed amphetamine salt has been approved for children age 3 + and methylphenidate has been used in FDA funded studies on preschool children; American Pediatric Association guidelines are also recommend for the preschool children) and these are the age ranges where children are most likely to present for treatment of irritability.

2. Meets diagnostic criteria for any presentation type of ADHD. ADHD status will be assessed on the NIMH Computerized Diagnostic Interview Schedule for Children (C-DISC).54 The C-DISC will also be used to assess psychiatric comorbidity, with diagnoses confirmed by an MD/PhD prior to eligibility decisions. Symptom severity for ADHD, irritability and Oppositional Defiant Disorder (ODD) will be assessed using the Disruptive Behavior Disorders (DBD) Parent Rating Scale which is similar to the Vanderbilt, rating symptoms on a 0-3 likert.24 In accordance with previous studies of irritability in ADHD, the DBD irritability score (range 0-9) will be the primary outcome, with a moderate level of irritability (≥5) required for entry.12 DMDD status will be assessed using Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (KSADS-PL) but DMDD will not be required for entry as subthreshold levels of irritability produce significant impairment.7 3. Sex: male or female 4. Fluent in written and spoken English.

Exclusion Criteria:

1. Age <5 years of age or >12 years of age.
2. Children with significant visual or hearing deficits or sensitivity to loud noises as test performance requires intact hearing and vision.
3. Children with a latex allergy as the sensors used in electrophysiology assessments have a latex component.
4. Serious neurological conditions that impacts cognition, such as an active seizure disorder
5. Current psychotropics other than FDA approved ADHD medications, as medication will be withheld on testing days. Unlike most other psychotropic medications, CNS stimulants can be withheld for brief periods and acutely restarted with no safety risks and lengthy titration process. Numerous ADHD studies have safely withdrawn these medications or substituted inert placebo for testing or clinical observation. Children taking an approved nonstimulant for ADHD plus a CNS Stimulant medication will be allowed to participate and will just have their CNS stimulant dose withheld on testing days.
6. Prominent traits of autism spectrum disorder (Social Communication Questionnaire Score >15), marked developmental delay or psychiatric conditions requiring urgent treatment (mania, psychoses, suicidal ideation).
7. Parent or child not fluent in English

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raman Baweja, MD, MS, Principal Investigator — Penn State Health
Locations (1):
- Penn State Hershey, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medication Arm
Started | 11
Completed | 9
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Medication Arm
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 8 [5 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Parent Rated Irritability on the IOWA Connor Irritability Score From Baseline to 6 Weeks.
Description: The primary outcome in this study was that change in parent rated irritability on the IOWA Connor irritability score. Parent Rating Scale rating symptoms on a 0-3 likert. Higher scores mean severe symptoms This scales has 3 items, which are reported as Not at all (0), just a little (1), pretty much (2) and very much (3) Total score is calculated by summiting all items. Total Score Ranges (0-9), higher score indicates more irritability.
Time Frame: Baseline and 6 weeks
Population: Nine patients completed the study. However, data for this outcome was missing for one patient, so the outcome was analyzed for eight patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Arm
Number analyzed (Participants) | 8
score on a scale | 3.13 (2.53)

2. Primary Outcome: Change in Parent-rated ADHD Symptoms, as Measured by the IOWA Conners Score, From Baseline to 6 Weeks.
Description: Symptom severity for ADHD symptoms will be assessed using the IOWA Connor Parent Rating Scale rating symptoms on a 0-3 likert. Higher scores mean severe symptoms This scale has 5 items, which are reported as Not at all (0), just a little (1), pretty much (2) and very much (3) Total score is calculated by summiting all items. Total Score Ranges (0-15). higher score indication of more ADHD symptoms.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Arm
Number analyzed (Participants) | 8
score on a scale | 4.38 (2.14)

3. Primary Outcome: Change in Parent-rated ODD Symptoms, as Measured by the IOWA Conners Score, From Baseline to 6 Weeks.
Description: Oppositional Defiant Disorder (ODD) symptoms were assessed using the IOWA Connor Parent Rating Scale rating symptoms on a 0-3 likert. Higher scores mean severe symptoms This scale has 5 items, which are reported as Not at all (0), just a little (1), pretty much (2) and very much (3) Total score is calculated by summiting all items. Total Score Ranges (0-15). Higher scores reflect greater levels ODD symptoms
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Arm
Number analyzed (Participants) | 8
score on a scale | 3.88 (4.12)

4. Secondary Outcome: Change in Parent-rated Impairment, as Measured by the Impairment Rating Scale (IRS), From Baseline to 6 Weeks.
Description: Parents completed the Impairment Rating Scale (IRS) to assess functioning across multiple domains. The IRS evaluates impairment in peer relationships, interactions with siblings and parents, academic performance, classroom behavior, self-esteem, family functioning, and overall functioning. Each item is rated on a 0-6 scale, and a total score is calculated by summing all item scores. Total scores range from 0 to 48, with higher scores indicating greater impairment.
Time Frame: Baseline and 6 weeks
Population: Nine patients completed the study. However, data for this variable was missing for one patient, so the outcome was analyzed for eight patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Arm
Number analyzed (Participants) | 8
score on a scale | 14.56 (6.53)

5. Secondary Outcome: Modified Overt Aggression Scale (MOAS)
Description: Parents completed the Modified Overt Aggression Scale (MOAS) to measure aggression. The Modified Overt Aggression Scale (MOAS) is a structured 20-item assessment tool used to measure the frequency and severity of aggressive behaviors. It categorizes aggression into four domains: verbal aggression, aggression against property, aggression towards self-directed, and physical aggression against others. Each item is rated on a scale from 0 (no aggression) to 4 (severe aggression), and scores within each domain are weighted (Verbal = ×1, Property = ×2, Autoaggression = ×3, Physical = ×4) to calculate a total weighted score ranging from 0 to 100. Higher scores indicate greater overall aggression.
Time Frame: Baseline
Population: All 11 participants at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Arm
Number analyzed (Participants) | 11
score on a scale | 28.27 (28.78)

6. Secondary Outcome: Inventory of Callous Unemotional Traits
Description: Parents completed Inventory of Callous Unemotional Traits to measure callous-unemotional characteristics. The Inventory of Callous-Unemotional Traits (ICU) is a 24-item scale designed to assess callous-unemotional traits in youth. Each item is rated on a 4-point scale ranging from 0 (Not at all) to 3 (Definitely true), producing a total score between 0 and 96. Higher scores reflect increased levels of callous-unemotional characteristics.
Time Frame: Baseline
Population: All 11 participants at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Arm
Number analyzed (Participants) | 11
score on a scale | 26 (5.06)

7. Secondary Outcome: Change in Parent-rated Affective Reactivity Index Total Score, as Measured by the Affective Reactivity Index, From Baseline to 6 Weeks.
Description: Parents completed the Affective Reactivity Index as an additional measure of irritability. The Affective Reactivity Index (ARI) is a 7-item scale used to assess irritability in youth. Each item is rated on a 3-point scale, ranging from 0 (Not true) to 2 (Certainly true), resulting in a total score between 0 and 14. Higher scores reflect greater levels of irritability.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Arm
Number analyzed (Participants) | 8
score on a scale | 7.6 (1.68)

8. Secondary Outcome: Change in Parent-rated Side Effects, as Measured by the Pittsburgh Side Effects Rating Scale (PSERS), From Baseline to 6 Weeks
Description: Parents completed the Pittsburgh Side Effects Rating Scale (PSERS) to evaluate side effects. The Pittsburgh Side Effects Rating Scale (PSERS) is a tool used to assess side effects commonly associated with medication treatment for ADHD. It includes 13 items rated on a Likert scale ranging from 0 (None) to 3 (Severe), yielding a total score from 0 to 39. Higher scores indicate more severe side effects.
Time Frame: Baseline and 6 weeks
Population: Nine patients completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Arm
Number analyzed (Participants) | 9
score on a scale | 1 (3.32)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: A total of 11 patients were enrolled in the study. Two patients dropped out following the baseline assessment and did not initiate study medication. Therefore, adverse event outcomes were reported for the remaining nine participants who received the intervention.
Arm/Group | Medication Arm
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT03279952/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT03279952/ICF_001.pdf